CLINICAL TRIAL: NCT02989051
Title: Fluids in Mechanically Ventilated Children With Acute Infectious Lung Disease: How Dry Should They be?
Brief Title: Fluid Restriction Keeps Children Dry
Acronym: LESSER
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, J.B.M. van Woensel, Professor, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016_096
Record Dates: First submitted 2016-12-05; First posted 2016-12-12 (Estimated); Last update posted 2016-12-12 (Estimated); Status verified 2016-12

CONDITIONS: Respiratory Infection; Fluid Overload; Critical Illness; Respiratory Insufficiency
MeSH Terms: conditions — Respiratory Tract Infections; Edema; Critical Illness; Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Restrictive fluid treatment (Experimental): Restrictive fluid regimen
  Interventions: Other: Restrictive fluid regimen
- Liberal fluid treatment (Active Comparator): This is seen as current standard clinical treatment, wherein patients will receive a more liberal fluid regimen.
  Interventions: Other: Liberal fluid regimen

INTERVENTIONS:
Other: Restrictive fluid regimen — In this treatment arm, patients will receive a maximal daily fluid intake of 70% of normal requirements (for a healthy child).
  Arms: Restrictive fluid treatment
Other: Liberal fluid regimen — This is considered current standard clinical treatment, wherein patients will receive a fluid regimen of >85% of normal fluid recommendations (for a healthy child).
  Arms: Liberal fluid treatment

SUMMARY:
Rationale: Fluid overload is a common complication in children who are admitted to the pediatric intensive care for mechanical ventilation. Acute lung infection is a frequent cause for admission to the PICU and forms an uniform group with a single organ failure. In these critically ill children, fluid overload is associated with adverse outcome. Restricting the volume of fluids already in an early stage of ICU admission may prevent fluid overload during mechanical ventilation and thus improve clinical outcome. However, at the same time fluid restriction may interfere with appropriate energy and macronutrient intake that is needed for recovery.

Objective: The main goal of this pilot study is to evaluate the feasibility of a restrictive fluid management protocol and investigate its effect on the occurrence of fluid overload in mechanically ventilated children with acute infectious lung disease.

Study design: Single-center prospective randomized feasibility and pilot study in preparation of a multi-center randomized controlled trial (RCT).

Study population: Mechanically ventilated children with (suspicion of) acute infectious lung disease admitted to the pediatric intensive care unit (PICU) of the Emma Children's Hospital, Academic Medical Center, Amsterdam.

Intervention: Patients receive either liberal (control group) or a restrictive (experimental group) fluid treatment, while ensuring appropriate caloric intake.

Main study parameters/endpoints: Primary outcomes are cumulative fluid balance and body weight during the first week of mechanical ventilation. Secondary outcomes (in preparation of the larger multi-center RCT) include: mortality, duration of mechanical ventilation and oxygenation indices. To determine the feasibility, in- and exclusion rate, adherence to treatment arms, need for fluid bolus, need for diuretics and hemodynamic indices as well as energy and protein intake are studied.

Both fluid management protocols reflect a variant of current clinical practice, hence will not provide extra burden or risk to patients included in the study. Patients will be randomized to either of the fluid protocol arms on admission to the PICU (at start of mechanical ventilation). Patients included in the restrictive fluid treatment arm might have direct benefit from the study if indeed fluid overload is less common in this group.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent by parents or legal caretakers
* Admitted to the PICU of the Emma Children's Hospital, Academic Medical Center, Amsterdam, The Netherlands
* Intubated and mechanically ventilated, with an anticipated duration of mechanical ventilation of at least 72 hours at enrolment (as judged by investigator or pediatrician on duty)
* Patients with an acute infectious lung disease, including (suspected) viral, bacterial or fungal infection

Exclusion Criteria:

* Patients in need of a particular fluid regimen (either restrictive or liberal) due to their medical history (e.g. cardiovascular disease and/or congenital (cyanotic) heart disease)
* Use of previous and/or maintenance diuretic treatment
* Ongoing (fluid) resuscitation on admission
* Acute kidney injury with need for renal replacement therapy

Ages: 1 Week to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-09 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Cumulative fluid balance | First week of mechanical ventilation
Body weight | First week of mechanical ventilation

SECONDARY OUTCOMES:
Duration of mechanical ventilation | Through study completion, an average of 1 week
Oxygenation indices | Through study completion, an average of 1 week
Mortality | Up to 90 days after admission

OTHER OUTCOMES:
In- and exclusion rate | Through study completion, an average of 1 week
Adherence to treatment arms | Through study completion, an average of 1 week
Need for fluid bolus | Through study completion, an average of 1 week
Need for diuretics | Through study completion, an average of 1 week
Need for vasopressors or inotropic drugs | Through study completion, an average of 1 week
Energy and protein intake | Through study completion, an average of 1 week
Gastrointestinal complaints | Through study completion, an average of 1 week
Hemodynamic indices | Through study completion, an average of 1 week
Occurrence of electrolyte imbalances | Through study completion, an average of 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- Academic Medical Center, Amsterdam, Netherlands

REFERENCES:
- [Derived] Ingelse SA, Geukers VG, Dijsselhof ME, Lemson J, Bem RA, van Woensel JB. Less Is More?-A Feasibility Study of Fluid Strategy in Critically Ill Children With Acute Respiratory Tract Infection. Front Pediatr. 2019 Dec 10;7:496. doi: 10.3389/fped.2019.00496. eCollection 2019. PMID 31921715